CLINICAL TRIAL: NCT04542993
Title: Can SARS-CoV-2 Viral Shedding in COVID-19 Disease be Reduced by Resveratrol-assisted Zinc Ingestion, a Direct Inhibitor of SARS-CoV-2-RNA Polymerase? A Single Blinded Phase II Protocol (Reszinate Trial)
Brief Title: Can SARS-CoV-2 Viral Load and COVID-19 Disease Severity be Reduced by Resveratrol-assisted Zinc Therapy
Acronym: Reszinate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty accruing patients
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: SHS KAPH NSWE 20090
Record Dates: First submitted 2020-09-08; First posted 2020-09-09 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: covid19; SARS-CoV-2; zinc; resveratrol
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — picolinic acid; Resveratrol

STUDY DESIGN:
Intervention Model Description: Placebo controlled Resveratrol and Zinc combination therapy
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol and Zinc Picolinate combination therapy (Active Comparator): Resveratrol and Zinc Picolinate combination therapy
  Interventions: Dietary Supplement: Zinc Picolinate; Dietary Supplement: Resveratrol
- Resveratrol Placebo and Zinc Placebo combination therapy (Placebo Comparator): Placebo Resveratrol and Placebo Zinc combination therapy
  Interventions: Dietary Supplement: Zinc Picolinate Placebo; Dietary Supplement: Resveratrol Placebo

INTERVENTIONS:
Dietary Supplement: Zinc Picolinate — Zinc Picolinate (50 mg PO TID x 5 days)
  Arms: Resveratrol and Zinc Picolinate combination therapy
Dietary Supplement: Resveratrol — Resveratrol 2 grams po BID x 5 days
  Arms: Resveratrol and Zinc Picolinate combination therapy
Dietary Supplement: Zinc Picolinate Placebo — Zinc Picolinate Matched Placebo PO TID x 5 days
  Arms: Resveratrol Placebo and Zinc Placebo combination therapy
Dietary Supplement: Resveratrol Placebo — Resveratrol Matched Placebo PO BID x 5 days
  Arms: Resveratrol Placebo and Zinc Placebo combination therapy

SUMMARY:
Administration of Zinc and resveratrol or double placebo for a period of 5 days and will be monitored for a 14 day period in covid-19 positive patients in an outpatient setting

DETAILED DESCRIPTION:
Research Question: In ambulatory, non-hospitalized patients with SARS-CoV-2 infection, is it possible to utilize resveratrol as a transporter for zinc treatment as means to minimize viral load and severity of resulting COVID-19 disease?

60 ambulatory SARS-CoV-2 positive volunteers who will be randomized into one of two treatment arms to receive either Zinc and resveratrol or double placebo for a period of 5 days and will be monitored for a 14 day period. It is anticipated to take approximately 20 weeks to accrue this cohort resulting in an estimated active project period of 22 weeks, although it may take up to 12 additional weeks to collect all of the data related to COVID-19 admissions in the cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 - 75) with a nasal swab confirmed SARS-CoV-2 infection; testing positive within 4 days of enrollment
2. Ability to read, understand and provide informed consent (no legally authorized representatives may consent on their behalf) and study assessments in English
3. Ability for subject to comply with the requirements of the study (must/will have a valid email address, internet connection and phone number)
4. Willingness to self limit medications and supplements and report what they are taking
5. Comfortable self-administering oral medication and nasal swab sampling
6. Willingness to permit a review of their medical history and to provide medical data from their electronic medical record for the period of enrollment (14 days) and until resolution of Covid-19 related events. Individuals who are not current Swedish patients will be asked to identify their provider of record and provide access to specific elements of their electronic health record.
7. Reside within twenty-five miles of one of the Swedish campuses: First Hill, Ballard, Edmonds, Issaquah, Cherry Hill.

Exclusion Criteria:

1. Reported history or evidence of impaired liver or kidney function: GFR <30 or bilirubin >2x ULT or INR > 2x ULT in the absence of anticoagulants
2. Known hypersensitivity to zinc or resveratrol
3. Diagnosis of COVID-19 or SARS-CoV-2 infection >4 days before enrollment
4. Preexisting severe pulmonary disease requiring supplemental oxygen
5. Clinically evident impairment of cognitive function, per physician discretion
6. Active substance abuse that may prevent the subject from completing the protocol requirements, per physician discretion.
7. Active psychotic or affective disorder that may prevent the subject from completing the protocol requirements, per physician discretion.
8. Pregnant or lactating females.
9. Coumadin treatment that can not be halted during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Reduction in SARS-CoV-2 Viral load | 1 year
  Viral AUCs normalized to peak viral load and housekeeper genes will be calculated, the AUCs on subjects with complete data will be used as dependent measures in t-tests, regressions and repeated measures mixed ANOVAs to compare viral load reduction between groups
Reduction in Severity of COVID-19 Disease | 1 year
  Review of healthcare resource utilization during study period

CONTACTS AND LOCATIONS:
Overall Officials: Hank Kaplan, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Currently no plan to make IPD available